CLINICAL TRIAL: NCT06125379
Title: Investigating the Effectiveness of Mindfulness-based Intervention on Teachers' Stress and Psychological Well-being in Rural Indonesia
Brief Title: Brief Mindfulness-based Intervention for Indonesian Teacher in Rural Area
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University Malaysia (Other)
Collaborators: Universitas Ahmad Dahlan (Other)
Responsible Party: Principal Investigator, Jamilah Hanum Abdul Khaiyom, PhD, Principal Investigator, International Islamic University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012211183
Record Dates: First submitted 2023-09-26; First posted 2023-11-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Stress, Psychological
Keywords: mindfulness; teacher; Indonesia; perceived stress; well-being
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MindCARE (Experimental): Group A is an experimental group that will receive mindfulness intervention for 4 consecutive weeks. Group A consists of 2-3 cohorts with 10-15 subjects per cohort.
  Interventions: Behavioral: brief mindfulness
- Wait-list control group (No Intervention): Group B is the wait-list control group which did not receive any intervention for 4 weeks.

INTERVENTIONS:
Behavioral: brief mindfulness — The mindfulness intervention protocol in this study is an adaptation of the Mindfulness Based Stress Reduction (MBSR) protocol with the cultural adaptation suits Indonesia population with addition of Islamic elements (i.e., a series of spiritual approaches) to improve emotional regulation, make sense of their life, be grateful and feel closer to God.
  Other Names: MindCARE (Mindfulness for Compassion and Relieve Stress)
  Arms: MindCARE

SUMMARY:
A randomized controlled trial to assess the effectiveness of the brief mindfulness on teachers' perceived stress and their psychological well-being.

DETAILED DESCRIPTION:
Teacher in early childhood education (ECE) in Indonesia is experiencing high intense stress due to work environment, class management, child behaviour problem, and lack administrative support. Stress has also shown negatively impact their psychological well-being, quality of teaching, and to children's' executive function. Research about stress and the effects on teacher well-being is especially lacking for rural schools. They represent a forgotten minority and thus, teacher from rural area need a prompt and direct support in terms of stress management strategies.

This study employs a randomized wait-list controlled trial design (RCT) with an assessment before and after treatment. 4-weeks brief mindfulness-based protocol will be given to 40 teachers as experimental group. 40 other teachers receive wait-list treatment will assign as control group. Measurement of perceived stress level will be using Indonesian version of Perceived Stress Scale (PSS), psychological wellbeing will be measure using Indonesian Well-being Scale (IWS), and mindfulness traits will be measure using Indonesian version of Five Factor Mindfulness Questionnaire (FFMQ). Data analysis using MANOVA and ANOVA to measure the differences between groups and within groups for all tests and constructs measured.

ELIGIBILITY:
Inclusion Criteria:

* minimum two years of work experience as early childhood education teacher.
* minimum 25 years of age.
* scoring Moderate (total score 14-26) to High (total score 27-40) perceived stress on PSS-10

Exclusion Criteria:

* have received any formal / manualized mindfulness training prior.
* have ever been diagnosed with chronic stress or other related mental disorders such as anxiety, depression, PTSD.
* people with a history or tendency to commit suicide.
* people with addictive substance dependence who are recovering less than one year.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS | 4 weeks
  The Perceived Stress Scale (PSS-10) is a 10-item questionnaire widely used to assess stress levels in young people and adults aged 12 and above. It evaluates the degree to which an individual has perceived life as unpredictable, uncontrollable and overloading over the previous month. The PSS score is obtained by summing across all items. A total PSS-10 score from 0 to 40 is presented, with higher scores representing higher levels of stress.

SECONDARY OUTCOMES:
Indonesian Well-being Scale (IWS) | 4 weeks
  The IWS is a well-being self-report instrument developed for the Indonesian general population. The scale consisted of 20 favourable items asking the respondent's sense of well-being in five different domains; Basic Needs (BN), Social Relation (SN), Acceptance (SA), Gratitude (GR), and Spirituality (SP). Score is ranging from 20 (minimum) to 100 (maximum), with higher score indicate higer psychological well-being.
Five Facet Mindfulness Scale (FFMQ) | 4 weeks
  The FFMQ consists of 39 items asking the individual to rate the extent to which a statement pertaining to mindfulness is applicable, on a scale from 1(never or rarely true) to 5 (very often or always true). Obtained score ranging from 39 (minimum) to 195 (maximum). Nineteen of the 39 items are reverse scored. These 19 items were reverse-scored prior to analysis, such that higher scores indicate higher mindfulness. Seven of the items comprise the non-reactivity facet, and eight items comprise each of the observing, describing, acting with awareness, and non-judging facets. Total scores for each facet are computed by summing the items after reverse scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Jamilah HA Khaiyom, Doctoral, Principal Investigator — International Islamic University
Locations (1):
- Ahmad Dahlan University, Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT06125379/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT06125379/ICF_001.pdf